CLINICAL TRIAL: NCT05662891
Title: The Effect of Blood Flow Restriction Applied During Nordic Hamstring Exercise on Neuromuscular Activation and Endothelial Function
Brief Title: The Effect of Blood Flow Restriction Applied During Nordic Hamstring Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fuat YÜKSEL, Dr./ Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-77082166-604.01.02-18938
Record Dates: First submitted 2022-11-24; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Endothelial Dysfunction; Hamstring Injury
Keywords: blood flow restriction; nordic hamstring exercise; endothelial function; muscular activation
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled single-blind study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction + Nordic hamstring exercise (Experimental)
  Interventions: Other: Blood Flow Restriction
- Nordic hamstring exercise (Experimental)
  Interventions: Other: Blood Flow Restriction

INTERVENTIONS:
Other: Blood Flow Restriction — After randomization, a cuff was placed proximal to one lower extremity. Blood flow was restricted from 60% of the arterial occlusion pressure. The other extremity was determined as the control group. 3x5 nordic hamstring exercises were performed. Surface emg was measured for hamstring muscles during exercise.
  Other Names: Nordic Hamstring Exercise

SUMMARY:
The aim of this study is to investigate the effects of blood flow restriction applied during nordic hamstring exercise on neuromuscular activation and endothelial function.

ELIGIBILITY:
Inclusion Criteria: Ankle arm index above 0.9

-

Exclusion Criteria:

* Having chronic diseases such as coronary heart disease, kidney diseases, diabetes, uncontrollable hypertension
* Having a history of deep vein thrombosis
* Having a previous hamstring injury
* To smoke
* Having a Body Mass Index over 25
* Having a history of major surgery

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function | It was evaluated for the control and experimental extremities before exercise.
  Endothelial function was evaluated with flow-mediated dilation.
Surface EMG | During exercise
  It was evaluated for the biceps femoris and semitendinosus muscles of the control and experimental extremities during Nordic hamstring exercise.
Endothelial function | It was evaluated for the control and experimental extremities 15 minutes after exercise. ( Outcomes were evaluated as acute.)
  Endothelial function was evaluated with flow-mediated dilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No